CLINICAL TRIAL: NCT03744819
Title: Exploration of Potential Biomarkers to Predict Tumor Response to Radiotherapy in Patients With Solid Tumors
Brief Title: Biomarkers for Prediction of Tumor Response to Radiotherapy
Status: Recruiting | Type: Observational
Sponsor: Chuangzhen Chen (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor-Investigator, Chuangzhen Chen, Deputy Director, Department of Radiation Oncology, Shantou University Medical College
Organization: Shantou University Medical College (Other)
Other Study IDs: IMRM2018
Record Dates: First submitted 2018-11-04; First posted 2018-11-16 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor samples, peripheral blood and microbiota
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to explore potential biomarkers for prediction of therapeutic outcomes in patients with solid tumors after radiotherapy

DETAILED DESCRIPTION:
Patients pathologically confirmed with solid tumors that requires radiotherapy or surgery will be recruited to this study. Tumor samples were obtained from patients underwent surgery to establish the baseline status of biomarker assessed. Peripheral and microbiota will also be collected before and after surgery. For patients undergoing radiotherapy, tumor biopsy as well as collection of blood samples and microbiota will be performed during the course of treatment. These biological specimens will be used for assessment of tumor phenotypes and for exploration of potential biomarkers that could predict the tumor response to therapeutics and prognsis in patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Pathological proven diagnosis of solid tumors
* Tumor accessible for biopsy during the course of radiotherapy or tumor samples could be obtained via surgery
* Patient must provide study-specific informed consent prior to study entry

Exclusion Criteria:

* History of autoimmune diseases
* History of immunotherapy
* Prior radiation therapy that would result in overlap of planned radiation therapy fields
* Will receive immunotherapy during the course of radiotherapy
* Contraindications for biopsy, such as high bleeding risk

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients proven diagnosis of solid tumors and will have radiotherapy as part of their therapeutic regimens or will undergo surgery in Cancer Hospital of Shantou University Medical College.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-10-29 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Expression status of biomarkers and their dynamic changes during treatment and follow-up | From the date of enrollment until the date of disease progression, assessed up to 3 years
  Expression status of biomarkers and their dynamic changes in patients' biological specimens through the course of treatment and during follow-up as assessed by a variety of means, including RNA-seq, DNA-seq, RT-qPCR, IHC, WB and ELISA.
Tumor short-term response to therapeutics | Within 1 month after the completion of radiotherapy
  For patients treated with radiotherapy, shortly after the completion of treatment, the short-term response was assessed by using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST1.1) .
Tumor long-term response to therapeutics | up to 3 years of follow-up
  For patients treated with radiotherapy, tumor response was assessed by using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST1.1) .

SECONDARY OUTCOMES:
Disease-specific survival | up to 3 years of follow-up
  The tumor disease-specific survival of patients

OTHER OUTCOMES:
Overall survival | up to 3 years of follow-up
  The overall survival of patients

CONTACTS AND LOCATIONS:
Overall Officials: Chuangzhen Chen, MD, Principal Investigator — Affiliated Cancer Hospital of Shantou University Medical College
Locations (1):
- Cancer Hospital, Shantou University Medical College, Shantou, Guangdong, China